CLINICAL TRIAL: NCT02616614
Title: Multicenter, Double-blind, Randomized, Parallel-group, Placebo-controlled Study to Evaluate the Bioequivalence of a Generic Clindamycin 1.2% and Benzoyl Peroxide 3.75% Gel to Onexton® Gel in Subjects With Acne Vulgaris
Brief Title: Double-blind Placebo-controlled Trial of Generic Clindamycin/Benzoyl Peroxide Gel Versus Onexton Gel in Acne Vulgaris
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Actavis Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: WAT/CMBP/2015
Record Dates: First submitted 2015-11-25; First posted 2015-11-30 (Estimated); Results first posted 2020-05-27 (Actual); Last update posted 2020-05-27 (Actual); Status verified 2020-05

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — clindamycin phosphate benzoyl peroxide combination; Clindamycin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Onexton gel (Active Comparator): Clindamycin 1.2% and benzoyl peroxide 3.75% topical gel Applied a thin film of medication onto 6 areas of the face (chin, left cheek, right cheek, nose, left forehead, and right forehead) once daily
  Interventions: Drug: Onexton
- Clindamycin/benzoyl peroxide gel (Experimental): Generic clindamycin 1.2% and benzoyl peroxide 3.75% topical gel. Applied a thin film of medication onto 6 areas of the face (chin, left cheek, right cheek, nose, left forehead, and right forehead) once daily
  Interventions: Drug: Clindamycin/benzoyl peroxide gel
- Placebo (Placebo Comparator): A vehicle gel. Applied a thin film of medication onto 6 areas of the face (chin, left cheek, right cheek, nose, left forehead, and right forehead) once daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Onexton — Topical gel for treating acne
  Other Names: Clindamycin/benzoyl peroxide gel
  Arms: Onexton gel
Drug: Clindamycin/benzoyl peroxide gel — Generic Clindamycin/benzoyl peroxide gel for treating acne
  Other Names: Clindamcyin Phosphate; BPO
  Arms: Clindamycin/benzoyl peroxide gel
Drug: Placebo — Vehicle gel used as a placebo
  Other Names: Vehicle
  Arms: Placebo

SUMMARY:
Actavis has developed a generic formulation of clindamycin 1.2% and benzoyl peroxide 3.75% gel. This study is designed to evaluate the safety and efficacy of this formulation in subjects with Acne Vulgaris

DETAILED DESCRIPTION:
This is a randomized, double blind, three-arm, parallel group, placebo control bioequivalence study with clinical endpoint, at multiple study sites, designed to establish bioequivalence of clindamycin 1.2% and benzoyl peroxide 3.75% gel of Actavis and Onexton® (clindamycin 1.2% and benzoyl peroxide 3.75%) gel in the treatment of subjects with Acne Vulgaris.

The primary objective is to evaluate the bioequivalence of a generic of clindamycin 1.2% and benzoyl peroxide 3.75% gel to Onexton® in the treatment of subjects with acne vulgaris.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or non-pregnant female aged ≥ 12 and ≤ 40 years with a clinical diagnosis of acne vulgaris
* On the face, ≥25 non-inflammatory lesions (i.e., open and closed comedones) and ≥ 20 inflammatory lesions (i.e., papules and pustules) and ≤ 2 nodulocystic lesions (i.e., nodules and cysts). For the purposes of study treatment and evaluation, these lesions should be limited to the facial treatment area. Counts of nodules and cysts should be reported separately and not included in the inflammatory or non-inflammatory lesion counts. Lesions involving the eyes and scalp should be excluded from the count. (Subjects may have acne lesions on other areas of the body (e.g., on the back)).
* Subjects must have Investigator's Global Assessment (IGA) of acne severity grade 2, 3, or 4.
* Willing to refrain from use of all other topical acne medications or antibiotics during the 12 week treatment period. Subjects may use other topical acne treatments that do not have significant or measurable systemic absorption for treatment of acne of the back, shoulders and chest (e.g. benzoyl peroxide, salicylic acid).
* Subjects who are 18 years of age or older must have provided Institutional Review Board (IRB) approved written informed consent. Subjects who are at least 12 years of age and less than 18 years of age must have provided IRB approved written assent; this written assent must be accompanied by an IRB approved written informed consent from the subject's legally acceptable representative (i.e., parent or guardian). In addition, all subjects or their legally acceptable representatives (i.e., parent or guardian) must sign a Health Insurance Portability and Accountability Act (HIPAA) authorization, if applicable.
* Male subjects and Female subjects of childbearing potential must use accepted methods of birth control or must agree to practice abstinence, from study start to 30 days after the last administration of study drug. All female subjects are considered to be of childbearing potential unless they have been surgically sterilized or have been postmenopausal for at least 1 year. Any of the following methods of birth control are acceptable: oral contraceptives, contraceptive patches/implants (e.g., Norplant®), vaginal ring (NuvaRing®), Depo-Provera® (Medroxy progesterone acetate), double barrier methods (e.g., condom and spermicide) or intrauterine device (IUD).
* Female subjects of child bearing potential must have a negative urine pregnancy test at baseline.
* Subjects who use make-up must have used the same brands/types of make-up for a minimum period of 14 days prior to study entry and must agree to not change make-up brand/type or frequency of use throughout the study.

Exclusion Criteria:

* History of hypersensitivity or allergy to clindamycin or benzoyl peroxide and/or any of the study medication ingredients or lincomycin or any other allowed product used during the study.
* Presence of any skin condition that would interfere with the diagnosis or assessment of acne vulgaris (e.g., on the face: rosacea, dermatitis, psoriasis, squamous cell carcinoma, eczema, acneform eruptions caused by medications, steroid acne, steroid folliculitis, or bacterial folliculitis).
* Excessive facial hair (beards, sideburns, moustaches, etc.) that would interfere with diagnosis or assessment of acne vulgaris. Patient is allowed to shave the excessive facial hair at least a day before visiting the site for study assessments.
* Use within 6 months prior to baseline of oral retinoids (e.g. Accutane®) or therapeutic vitamin A supplements of greater than 10,000 units/day.
* Use for less than 3 months prior to baseline of estrogens or oral contraceptives; use of such therapy must remain constant throughout the study.
* Use on the face within 1 month prior to baseline or during the study of: 1) cryodestruction, 2) dermabrasion, 3) photodynamic therapy, 4) acne surgery, 5) intralesional steroids, or 6) x-ray therapy.
* Use within 1 month prior to baseline of: 1) spironolactone, 2) systemic steroids, 3) systemic antibiotics, 4) systemic treatment for acne vulgaris or 5) systemic anti-inflammatory agents.
* Use within 2 weeks prior to baseline of: 1) topical steroids, 2) topical retinoids, 3) topical acne treatments including over-the-counter preparations, 4) topical anti- inflammatory agents, 5) medicated cleansers or 6) topical antibiotics.
* Subjects who have acne fulminans, and secondary acne (e.g., chloracne and drug induced acne) will be excluded from participation.
* Female subjects who are pregnant, nursing or planning to become pregnant during study participation (Visit 1 through Visit 4 and 30 days post visit 4) will be excluded from study participation.
* Subjects who have received radiation therapy and/or anti-neoplastic agents within 90 days prior to baseline will be excluded from study participation.
* Subjects who have unstable medical disorders that are clinically significant or life-threatening diseases will be excluded from study participation.
* Subjects who have on-going malignancies requiring systemic treatment will be excluded from study participation. In addition, subjects who have any malignancy of the skin of the facial area will be excluded from study participation.
* Subjects who engage in activities that involve excessive or prolonged exposure to sunlight or weather extremes, such as wind or cold, will be excluded from study participation.
* Subjects who have facial sunburn will be excluded from study participation
* Subjects who consume excessive amounts of alcohol (greater than two drinks per day) or use drugs of abuse (including, but not limited to, cannabinoids and cocaine) as judged by their medical history will be excluded from study participation.
* History or presence of significant smoking (more than 10 cigarettes or any other form of tobacco smoking/day or consumption of tobacco products).
* Systolic blood pressure less than 90 mm Hg or more than 140 mm Hg, Diastolic blood pressure less than 60 mm Hg or more than 90 mm Hg and Pulse rate less than 50 beats/minute or more than 100 beats/minute.
* Subjects who have participated in an investigational drug study (i.e., subjects have been treated with an investigational drug) within 1 month prior to baseline will be excluded from study participation. Subjects who are participating in non- treatment studies such as observational studies or registry studies can be considered for inclusion.
* Major illness, as per investigator's discretion, during 3 months before screening.
* Subjects who have been previously enrolled in this study will be excluded from study participation.
* Subjects who have had laser therapy and electrodesiccation to the facial area within 180 days prior to study entry will be excluded from participation.
* Subjects who have had cosmetic procedures (e.g., facials) which may affect the efficacy and safety profile of the investigational product within 14 days prior to study entry will be excluded from participation.
* Subjects who have had general anesthesia for any reason and subjects who have received neuromuscular blocking agents within 14 days prior to study entry will be excluded from study participation.
* Subjects who have a baseline score of 3 (severe, marked/intense) as per the Application Site Reaction Scale (Section 5.2) will be excluded from participation.
* Any employees or staff of the research site are excluded from study participation.

Ages: 12 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 862 (Actual)
Dates: Start 2015-05; Primary Completion 2015-10 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Henry lau, PhD, Study Director — Actavis Inc.
Locations (17):
- United States (17):
  - Alliance Dermatology, Phoenix, Arizona
  - Estudy, Chula Vista, California
  - Estudy, La Mesa, California
  - Tampa Bay Medical Research, Clearwater, Florida
  - AMB Research Center, Miami, Florida
  - Meridian Clinical Research, Savannah, Georgia
  - Heartland Research Assoc, Augusta, Kansas
  - Heartland Research Assoc, Wichita, Kansas
  - Sundance Clinical Research, St Louis, Missouri
  - Meridian Clinical Research, Norfolk, Nebraska
  - Meridian Clinical Research, Omaha, Nebraska
  - Dermatology Consulting Services, High Point, North Carolina
  - Sterling Research Group, Cincinnati, Ohio
  - Discover Research, Beaumont, Texas
  - DiscoverResearch Inc, Bryan, Texas
  - Reseacr Across America, Dallas, Texas
  - Clinical Research Assoc. of Tidewater, Norfolk, Virginia

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The populations for this study included the Safety Population, the Per-Protocol Population (PP), and the modified Intent-to-Treat (mITT) Population.
Groups:
- Generic Clindamycin 1.2% and Benzoyl Peroxide 3.75% Gel; Onexton (Clindamycin 1.2% and Benzoyl Peroxide 3.75% Gel); Vehicle Gel: Subjects applied one pea-sized amount of the investigational product to the entire face 1 time each day for a period of 84 days.
Period: Overall Study
Arm/Group | Generic Clindamycin 1.2% and Benzoyl Peroxide 3.75% Gel | Onexton (Clindamycin 1.2% and Benzoyl Peroxide 3.75% Gel) | Vehicle Gel
Started | 347 | 345 | 170
Safety Population (Randomized participants who received the study drug) | 329 | 328 | 161
mITT Population (Randomized participants, received at least 1 dose of study drug and at least 1 post-baseline visit) | 325 | 325 | 160
PP Population (Randomized subjects, compliant with study drug, completed study) | 253 | 255 | 122
Completed | 282 | 285 | 141
Not Completed | 65 | 60 | 29
Not completed — Withdrawal by Subject | 10 | 5 | 6
Not completed — Physician Decision | 2 | 1 | 0
Not completed — Adverse Event | 1 | 4 | 1
Not completed — Protocol Violation | 0 | 3 | 1
Not completed — Prohibited Medication | 12 | 9 | 5
Not completed — More than 3 applications missed | 6 | 8 | 1
Not completed — Lost to Follow-up | 31 | 28 | 13
Not completed — Pregnancy | 2 | 0 | 1
Not completed — Other | 1 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Reference Onexton (Clindamycin 1.2% and Benzoyl Peroxide 3.75); Vehicle Gel: Subjects applied one pea-sized amount of the investigational product to the entire face 1 time each day for a period of 84 days.
- Total: Total of all reporting groups
Arm/Group | Generic Clindamycin 1.2% and Benzoyl Peroxide 3.75% Gel | Reference Onexton (Clindamycin 1.2% and Benzoyl Peroxide 3.75) | Vehicle Gel | Total
Number analyzed (Participants) | 329 | 328 | 161 | 818
Age, Continuous [Mean (Standard Deviation); unit: years] | 20.6 (7.56) | 20.4 (7.04) | 20.1 (6.92) | 20.4 (7.23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 204 | 217 | 105 | 526
  Male | 125 | 111 | 56 | 292
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 76 | 89 | 45 | 210
  Not Hispanic or Latino | 253 | 239 | 116 | 608
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Asian | 4 | 2 | 1 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 82 | 86 | 42 | 210
  White | 225 | 224 | 110 | 559
  More than one race | 18 | 15 | 8 | 41
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in the Inflammatory (Papules and Pustules) Lesion Counts
Description: Percent change from baseline to Week 12 (Day 84) in the inflammatory (papules and pustules) lesion count in PP Population.
Time Frame: 12 weeks
Population: Using the per-protocol population.
Measure: Mean (Standard Deviation); unit: percentage of change
Groups:
- Generic Clindamycin and Benzoyl Peroxide: Clindamycin 1.2% and Benzoyl Peroxide 3.75% gel (Actavis Laboratories SLC)
- Reference Onexton (Clindamycin and Benzoyl Peroxide): Onexton gel (Clindamycin 1.3% and Benzoyl Peroxide 3.75%) (Valeant Pharmaceuticals North America LLC)
- Vehicle Gel: Vehicle Gel: Placebo product
Arm/Group | Generic Clindamycin and Benzoyl Peroxide | Reference Onexton (Clindamycin and Benzoyl Peroxide) | Vehicle Gel
Number analyzed (Participants) | 253 | 255 | 122
percentage of change | -63.81 (36.791) | -67.56 (28.405) | -53.78 (40.138)
Statistical Analysis 1: Comparison: Generic Clindamycin and Benzoyl Peroxide vs Reference Onexton (Clindamycin and Benzoyl Peroxide); Test type: Equivalence — Bioequivalence was established if the 90% CI for the difference was contained within the interval [0.80,1.25] for the PP population; Mean Difference (Net) = 0.95, 90% CI 2-sided [0.88 to 1.03]
Statistical Analysis 2: Comparison: Generic Clindamycin and Benzoyl Peroxide; Test type: Superiority; p = 0.0001, ANOVA
Statistical Analysis 3: Comparison: Reference Onexton (Clindamycin and Benzoyl Peroxide); Test type: Superiority; p < 0.0001, ANOVA

2. Primary Outcome: Percent Change in the Non-Inflammatory (Open and Closed Comedomes) Lesion Counts
Description: One of the co-primary endpoints was the percent change from baseline to Week 12 (Day 84) in the non-inflammatory (open and closed comedones) lesion counts in PP Population.
Time Frame: 12 weeks
Population: Using the per-protocol population.
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Generic Clindamycin and Benzoyl Peroxide | Reference Onexton (Clindamycin and Benzoyl Peroxide) | Vehicle Gel
Number analyzed (Participants) | 253 | 255 | 122
percentage of change | -49.58 (40.747) | -49.50 (32.872) | -37.50 (40.261)
Statistical Analysis 1: Comparison: Generic Clindamycin and Benzoyl Peroxide vs Reference Onexton (Clindamycin and Benzoyl Peroxide); Test type: Equivalence — Bioequivalence was established if the 90% CI for the difference was contained within the interval [0.80, 1.25] for the PP population; Mean Difference (Net) = 1.00, 90% CI 2-sided [0.90 to 1.11]
Statistical Analysis 2: Comparison: Generic Clindamycin and Benzoyl Peroxide; Test type: Superiority; p = 0.0002, ANOVA
Statistical Analysis 3: Comparison: Reference Onexton (Clindamycin and Benzoyl Peroxide); Test type: Superiority; p = 0.0006, ANOVA

3. Secondary Outcome: Number of Subjects With Treatment Success at Week 12
Description: The secondary efficacy endpoint was the IGA score, expressed in terms of proportion of subjects with treatment success or failure at Week 12, where "success" was defined as an IGA score that was at least 2 grades less than the baseline assessment.
Time Frame: 12 weeks
Population: Using the PP population.
Measure: Number; unit: participants
Groups:
- Vehicle Gel: Vehicle of the test product (Actavis Laboratories SLC)
Arm/Group | Generic Clindamycin and Benzoyl Peroxide | Reference Onexton (Clindamycin and Benzoyl Peroxide) | Vehicle Gel
Number analyzed (Participants) | 253 | 255 | 122
participants
  Success | 54 | 60 | 13
  Failure | 199 | 195 | 109
Statistical Analysis 1: Comparison: Generic Clindamycin and Benzoyl Peroxide vs Reference Onexton (Clindamycin and Benzoyl Peroxide); Bioequivalence was established if the 90% CI for the difference was contained within the interval (-0.20, +0.20); Test type: Equivalence — Bioequivalence was established if the 90% CI for the difference was contained within the interval (-0.20, +0.20); Mean Difference (Net) = -0.022, 90% CI 2-sided [-0.087 to 0.043] — Equivalence was based on difference in the number of subjects with success. Bioequivalence was established if the 90% CI for the difference was contained within the interval (-0.20, +0.20)

ADVERSE EVENTS:
Time Frame: Baseline to 12 Weeks
Description: Adverse events were collected from participants who were randomized and received the study drug.
  Safety population assessment
Arm/Group | Generic Clindamycin 1.2% and Benzoyl Peroxide 3.75% Gel | Reference Onexton (Clindamycin 1.2% and Benzoyl Peroxide 3.75) | Vehicle Gel
All-Cause Mortality (participants affected / at risk) | 0/329 | 0/328 | 0/161
Serious Adverse Events (participants affected / at risk) | 4/329 | 0/328 | 0/161
Other Adverse Events (participants affected / at risk) | 197/329 | 211/328 | 92/161
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Generic Clindamycin 1.2% and Benzoyl Peroxide 3.75% Gel (N=329) | Reference Onexton (Clindamycin 1.2% and Benzoyl Peroxide 3.75) (N=328) | Vehicle Gel (N=161)
Bipolar disorder (Psychiatric disorders) | 1 | 0 | 0
Cranio-cerebral injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 — Closed head injury
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 — Spontaneous abortion
Allergy to arthropod sting (Immune system disorders) | 1 | 0 | 0 — Bee sting with acute allergic reaction, likely anaphlactoid
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Generic Clindamycin 1.2% and Benzoyl Peroxide 3.75% Gel (N=329) | Reference Onexton (Clindamycin 1.2% and Benzoyl Peroxide 3.75) (N=328) | Vehicle Gel (N=161)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0 | 0
Extrasystoles (Cardiac disorders) | 2 | 0 | 1
Sinus tachycardia (Cardiac disorders) | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 1
Goitre (Endocrine disorders) | 1 | 0 | 0
Eye irritation (Eye disorders) | 1 | 0 | 0
Eye pain (Eye disorders) | 1 | 0 | 0
Eye swelling (Eye disorders) | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0
Aphthous stomatitis (Gastrointestinal disorders) | 0 | 0 | 1
Dental caries (Gastrointestinal disorders) | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 0 | 2
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0
Toothache (Gastrointestinal disorders) | 2 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0
Application site dryness (General disorders) | 11 | 9 | 2
Application site erosion (General disorders) | 1 | 0 | 0
Application site erythema (General disorders) | 5 | 6 | 0
Application site irritation (General disorders) | 0 | 3 | 3
Application site oedema (General disorders) | 0 | 0 | 1
Application site pain (General disorders) | 4 | 4 | 1
Application site pruritus (General disorders) | 4 | 5 | 3
Chest pain (General disorders) | 0 | 1 | 0
Cyst (General disorders) | 0 | 1 | 0
Face oedema (General disorders) | 3 | 5 | 2
Facial pain (General disorders) | 16 | 17 | 5
Inflammation (General disorders) | 0 | 1 | 0
Local swelling (General disorders) | 0 | 1 | 0
Oedema (General disorders) | 2 | 0 | 1
Pain (General disorders) | 8 | 3 | 0
Pyrexia (General disorders) | 1 | 0 | 0
Secretion discharge (General disorders) | 0 | 1 | 0
Non-alcoholic steatohepatitis (Hepatobiliary disorders) | 0 | 1 | 0
Allergy to arthropod sting (Immune system disorders) | 1 | 0 | 0
Body tinea (Infections and infestations) | 0 | 0 | 1
Breast abscess (Infections and infestations) | 0 | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0
Conjunctivitus (Infections and infestations) | 0 | 1 | 0
Gastroenteritis viral (Infections and infestations) | 2 | 0 | 0
Herpes simplex (Infections and infestations) | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 1 | 0
Kidney infection (Infections and infestations) | 0 | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 1 | 1
Oral herpes (Infections and infestations) | 0 | 0 | 1
Otitis media (Infections and infestations) | 0 | 1 | 0
Pharyngitis streptococcal (Infections and infestations) | 1 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0 | 0
Rash pustular (Infections and infestations) | 0 | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 1
Sinusitus (Infections and infestations) | 1 | 1 | 0
Skin infection (Infections and infestations) | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 3 | 2 | 0
Cartilage injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 1 | 0
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1 | 0
Joint injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 1 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Muscle strain (Injury, poisoning and procedural complications) | 1 | 1 | 1
Scar (Injury, poisoning and procedural complications) | 0 | 1 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 1 | 1 | 0
Sunburn (Injury, poisoning and procedural complications) | 1 | 4 | 1
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 1
Blood pressure increased (Investigations) | 0 | 1 | 0
Heart rate increased (Investigations) | 0 | 1 | 0
Heart rate irregular (Investigations) | 1 | 0 | 0
Investigation (Investigations) | 2 | 2 | 2
Investigation abnormal (Investigations) | 0 | 1 | 0
Weight increased (Investigations) | 1 | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Burning sensation (Nervous system disorders) | 0 | 0 | 1
Headache (Nervous system disorders) | 2 | 1 | 1
Migraine (Nervous system disorders) | 0 | 0 | 1
Paraesthesia (Nervous system disorders) | 2 | 1 | 1
Presyncope (Nervous system disorders) | 0 | 0 | 1
Sinus headache (Nervous system disorders) | 0 | 0 | 2
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0
Bipolar disorder (Psychiatric disorders) | 1 | 0 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 0 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 1 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
Acne (Skin and subcutaneous tissue disorders) | 9 | 9 | 10
Blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 127 | 138 | 56
Erythema (Skin and subcutaneous tissue disorders) | 55 | 58 | 31
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 2 | 2 | 1
Papule (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 59 | 70 | 31
Rash (Skin and subcutaneous tissue disorders) | 2 | 1 | 0
Scab (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Seborrhoea (Skin and subcutaneous tissue disorders) | 0 | 2 | 2
Skin burning sensation (Skin and subcutaneous tissue disorders) | 34 | 27 | 11
Skin erosion (Skin and subcutaneous tissue disorders) | 12 | 22 | 8
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 17 | 23 | 10
Skin swelling (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 5 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Artificial crown procedure (Surgical and medical procedures) | 0 | 1 | 0
Hot flush (Vascular disorders) | 0 | 0 | 1
Hypotension (Vascular disorders) | 1 | 4 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The results of the study may be published or presented by the Investigator(s) after the review by, and in consultation and agreement with the Sponsor, and such that confidential or proprietary information is not disclosed.